CLINICAL TRIAL: NCT02368925
Title: Clinical Trial to Evaluate Safety and Efficacy of Ultherapy™ System for Lifting Skin
Brief Title: Clinical Trial to Evaluate Safety and Efficacy of Ultherapy™ System for Lifting Skin on the Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-1411/274-002
Record Dates: First submitted 2015-02-15; First posted 2015-02-23 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Wrinkles
Keywords: Rhytids; Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy™ System (Experimental): Ultherapy™ System
  Interventions: Device: Ultherapy™ System

INTERVENTIONS:
Device: Ultherapy™ System — The Investigator will apply to the eligible subject the Study Device Ultherapy™ System with 200~260 lines of 3.0 and 4.5 probe respectively on the subject's neck.

SUMMARY:
Study is a prospective clinical trial to evaluate the efficacy of the Ulthera® System to improve Lifting Skin on the Neck. Changes from baseline in the FACE-Q Appraisal of Neck scale score and Global Aesthetic Improvement Scale scores will be assessed at study follow-up visits.

DETAILED DESCRIPTION:
Before Treatment:

The subject's eligibility (inclusion/exclusion criteria) will be assessed, and all subjects will check the FACE-Q Appraisal of Neck scale score

Treatment:

The Investigator will apply to the eligible subject the Study Device Ultherapy™ System with 200~260 lines of 3.0 and 4.5 probe respectively on the subject's neck.

Post-Treatment:

All subjects will visit the Institution at 12 weeks from the day of procedure, and will take photos of the neck. Efficacy evaluation will performed by the Photographic Evaluator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years.
* Subject in good health
* Subjects who desire improvement in neck skin

Exclusion Criteria:

* Presence of an active systemic infectious disease
* general disease or skin disorder in the area to be treated
* Pregnant or lactating subjects
* Previous episode of facial or neck surgery for wrinkle correction
* Subjects who have aesthetic addiction, drug abuse, alcohol abuse
* Subjects who were treated Botox or Filler at the neck area
* Subjects who had Auto-Immune disease

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Investigator Assessment of Improvement at 12 weeks post-treatment | 12 weeks post-treatment
  Investigator complete Global Aesthetic Improvement Scale at 12 weeks post-treatment by comparing subject's photographs

SECONDARY OUTCOMES:
Subject Assessment of Improvement at 12 weeks post-treatment | 12 weeks post-treatment
  Subjects complete a Patient Assessment Global Aesthetic Improvement Scale at 12 weeks posttreatment
Subjects' Assessment of Pain during treatment | Subjects were assessed for the duration of study treatment
  Pain score record using a Numeric Rating Scale (NRS,0-10) , with 0 representing no pain and 10 representing the worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: ChangSik Pak, Bachelor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No